CLINICAL TRIAL: NCT02000167
Title: Mitochondrial Dysfunction in Phelan-McDermid Syndrome: Explaining Clinical Variation and Providing a Path Towards Treatment
Brief Title: Mitochondrial Dysfunction in Phelan-McDermid Syndrome
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: St. Christopher's Hospital for Children (Other)
Responsible Party: Sponsor
Other Study IDs: 136271
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2015-06

CONDITIONS: Phelan-McDermid Syndrome
Keywords: Electron Transport Chain; Mitochondrial Disease; Chromosomal Deletion
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome; Mitochondrial Diseases; Chromosome Deletion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Phelan-McDermid Syndrome only: Diagnosed with Phelan-McDermid Syndrome; 50 subjects to be recruited. 1-21 years of age
- Co-morbid Phelan-McDermid Syndrome & Mitochodrial Disorder: 1-21 years of age; Diagnosed with Phelan-McDermid Syndrome AND diagnosed with Mitochondrial Disorder; 50 subjects to be recruited.

SUMMARY:
The purpose of this study is to determine whether a relationship exists between gene deletion(s) specific to the mitochondrial electron transport chain and presentation of clinical characteristics in patients with Phelan-McDermid Syndrome (PMS).

DETAILED DESCRIPTION:
Phelan-McDermid Syndrome (PMS) results from a deletion within the 22q13 chromosome region. Most children have specific physical morphology and developmental delays with many displaying characteristics of autism spectrum disorder (ASD) including abnormalities in social development. The behavioral aspect of PMS that parallels ASD has raised particular interest as the SHANK3 gene, which lies in the 22q13 region, is important for synaptic development, and animal SHANK3 knockout models demonstrate ASD characteristics thereby confirming the importance of this gene in PMS. However, despite the importance of the SHANK3 gene, individuals with PMS have variations in their development, behavior and medical characteristics that cannot be fully explained by the SHANK3 deletion.

Recently, Frye (2012) has noted the existence of 6 mitochondrial genes that lie slightly proximal to the SHANK3 gene within the 22q13 region. These include genes important electron transport change function (SCO2, NDUFA6), mitochondrial DNA (TYMP) and RNA (TRMU) metabolism, fatty acid metabolism (CPT1B) and tricarboxylic acid cycle function (ACO2). Since most Individuals with PMS have deletions that include chromosomal deletion outside of the SHANK3 region, it is very likely that many, if not most, of children with PMS may have deletions in these mitochondrial genes. Many of these genes have been linked to mitochondrial disease, even in the heterozygous state. Even if recognized, mitochondrial disease is only linked to a homozygous abnormal state (autosomal recessive), the loss of one gene (heterozygous state) could result in symptomatology when associated with deletions in other mitochondrial or non-mitochondrial genes. Abnormalities in mitochondrial pathways can result in neurologic and non-neurologic symptoms including those sometimes seen in children with PMS. Added with the SHANK3 deletion, abnormalities in these mitochondrial genes could explain variations in patterns of development and the eventual cognitive potential.

References: Frye RE. Mitochondrial disease in 22q13 duplication syndrome. J Child Neurol. 2012; 27(7):942-9.

ELIGIBILITY:
Inclusion Criteria:

* 1-21 years of age
* Diagnosed with Phelan-McDermid Syndrome AND diagnosed with Mitochondrial Disorder
* Diagnosed with Phelan-McDermid Syndrome

Exclusion Criteria:

* none

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be identified through the registry for this specific aim. PMS patients in the registry will be offered to be entered the study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Electron Transport Chain function derived from buccal cells of known PMS patients | Up to two years
  Electron transport chain (ETC) function will be measured in cells collected using Buccal swabs to determine if certain PMS patients symptomatology and clinical characteristics/variations can be explained due to variations in patterns of ETC function in this cohort

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, M.D./Ph.D., Principal Investigator — University of Arkansas for Medical Sciences; Arkansas Children's Hospital Research Institute; Michael J Goldenthal, Ph.D., Principal Investigator — Drexel University College of Medicine
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States